CLINICAL TRIAL: NCT02575690
Title: Effect of Spirulina Maxima Supplementation on Cardiovascular Risk in Obese Caucasians With Treated Hypertension:a Randomized Double-blind Placebo-controlled Study
Brief Title: Spirulina Supplementation and Cardiovascular Risk in Obese Caucasians With Treated Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pawel Bogdanski, Associate professor, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 599/12
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Obesity
Keywords: spirulina, placebo, obesity,antihypertensive treatment
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): Obese patients with well-treated hypertension that receive placebo (pure microcrystalline cellulose)
  Interventions: Other: Placebo
- Spirulina group (Experimental): Obese patients with well-treated hypertension that receive Hawaiian spirulina (Cyanotech Corporation, Hawaii, US)
  Interventions: Dietary Supplement: Spirulina

INTERVENTIONS:
Dietary Supplement: Spirulina — Individuals receive 2 g of spirulina daily, for 3 months.
  Arms: Spirulina group
Other: Placebo — Individuals receive a placebo daily, for 3 months.
  Arms: Placebo group

SUMMARY:
Potential protective cardiovascular effect of Spirulina maxima supplementation was studied in a double-blind placebo-controlled trial of obese subjects with treated hypertension, each randomized to receive spirulina or a placebo.

DETAILED DESCRIPTION:
Numerous publications have provided evidence of the effect of natural substances-supplements on improving endothelial function, and thus reducing the risk of cardiovascular diseases. Spirulina maxima (Arthrospira maxima) is a species of cyanobacterium, used as food additive because of its high levels of protein and essential nutrients, such as carotenoids, vitamins, and minerals. Various studies point to a possible beneficial effect of spirulina on the concentration of blood serum lipids and fasting glucose,body weight or blood pressure, however, the results of studies pertained to the effects of spirulina in individuals who, at the time of trial, were not taking medications. The aim of the study was to estimate an effect of Spirulina maxima supplementation on cardiovascular risk in obese Caucasians with treated hypertension. The anthropometric parameters, blood pressure, insulin sensitivity, plasma lipid levels, and stress oxidative biomarkers were measured at the baseline and after 3 months of supplementation with spirulina or placebo in the group of obese, hypertensive patients receiving standard antihypertensive treatment.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) equal to or greater than 30 kg/m2
* age 25 to 60 years
* stable body weight (< 3 kg self-reported change during the previous three months)
* well-controlled hypertension (meaning systolic blood pressure (SBP) less than 160 mmHg and/or diastolic blood pressure (DBP) less than 100 mmHg) with stable treatment for at least 6 months (the patients received one drug only)

Exclusion Criteria:

* secondary obesity or secondary hypertension
* diabetes
* a history of coronary artery disease
* stroke
* congestive heart failure
* malignancy
* a history of use of any dietary supplements within the three months prior to the study
* a current need for modification of antihypertensive therapy
* abnormal liver or kidney function
* any clinically significant process
* a history of infection in the month prior to the study
* nicotine or alcohol abuse
* or other condition that, in the opinion of the investigators, would make participation not in the best interest of the patient or could prevent, limit, or confound the protocol-specified efficacy assessments

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Body mass index | at baseline of the study

SECONDARY OUTCOMES:
blood pressure | At the baseline and following 3 months of treatment
Body mass index | 3 months
waist circumference | At the baseline and following 3 months of treatment
serum lipids | At the baseline and following 3 months of treatment
Total antioxidant status (TAS) evaluated by colorimetric method with Tas Randox kit | At the baseline and following 3 months of treatment
insulin estimated by immunoassay (DIAsource immunoassays) | At the baseline and following 3 months of treatment
interleukin-6 measured by an enzyme-linked immunosorbent assay (R&D Quantikine® Human Il-6 kit) | At the baseline and following 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Bogdanski, MD, PhD, Principal Investigator — Poznan University of Medical Sciences